CLINICAL TRIAL: NCT00724217
Title: The Effects of the Standard Process 21 Day Purification Program, on Serum Lipids, C-Reactive Protein, Homocystine, Blood Pressure, and Heart Rate Variability in Normal Weight and Overweight Participants Who Have Total Cholesterol Levels Over 180.
Brief Title: Standard Process 21 Day Purification Program Project
Acronym: SPPP
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Logan College of Chiropractic (Other)
Responsible Party: Rodger Tepe, PhD, Logan College of Chiropractic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RD0530080135
Record Dates: First submitted 2008-07-25; First posted 2008-07-29 (Estimated); Last update posted 2008-07-29 (Estimated); Status verified 2008-07

CONDITIONS: Hyperlipidemia
MeSH Terms: conditions — Hyperlipidemias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Normal weight (Experimental): BMI < 26
  Interventions: Other: Standard Process 21 Day Purification Program (SPPP)
- Overweight (Experimental): BMI >= 26
  Interventions: Other: Standard Process 21 Day Purification Program (SPPP)

INTERVENTIONS:
Other: Standard Process 21 Day Purification Program (SPPP) — The Standard Process 21 Day Purification Program (SPPP) consists of a controlled food intake regimen of mostly fruit and vegetables with restricted calories, protein and fats plus daily use of herbal and whole food based supplements.
  Arms: Normal weight
Other: Standard Process 21 Day Purification Program (SPPP) — The Standard Process 21 Day Purification Program (SPPP) consists of a controlled food intake regimen of mostly fruit and vegetables with restricted calories, protein and fats plus daily use of herbal and whole food based
  Arms: Overweight

SUMMARY:
To determine the effects of a commercially available dietary modification plus nutritional supplement regimen, the Standard Process 21 day Purification Program (SPPP), on serum lipids, C-reactive protein (CRP), homocysteine, body mass index (BMI), body weight, blood pressure, and heart rate variability (HRV) in normal weight (BMI < 26) and overweight (BMI 26 or above) participants who have total cholesterol levels over 180.

DETAILED DESCRIPTION:
Elevated low-density lipoprotein (LDL) cholesterol concentrations are a risk factor for cardiovascular diseases. (1) Cholesterol lowering drugs are the most frequently prescribed medications in the U.S. and are known to have muscle, kidney and liver side effects for some users. Recent reviews conclude that benefits outweigh risks reporting statin and other cholesterol-lowering drugs to be safe and effective for most users. (2, 3, 4, 5) The new blood cholesterol level guidelines may recommend that more people take cholesterol lowering medications. According to the American Heart Association (AHA), total cholesterol levels should be below 180 mg/dL, with levels from 200 mg/dL to 239 mg/dL considered borderline high. Total cholesterol of 240 mg/dL and above is considered high. (6) However, published studies on the effect of blood lipids suggested that the actual cholesterol level itself is not the most important risk factor. It is the ratio between the level of total cholesterol and HDL that played a major role in the cardiovascular risk. The ideal HDL/cholesterol ratio should be higher than 25%. The ideal triglyceride/cholesterol ratio should be below 2.0. It is estimated that over 50 million adults in the U.S. have lipid levels higher than the above recommendations. (6) For persons who prefer conservative care, dietary modification is considered a first approach to the treatment and control of high cholesterol. (1, 7, 8) Hypertension is another risk factor for cardiovascular diseases and has close links to high blood cholesterol. (8) Between 40 and 50 million Americans have hypertension, which is defined as systolic blood pressure of at least 140 mm Hg or diastolic blood pressure of at least 90 mm Hg. (8) Hypertension is strongly, continuously, and independently related to coronary artery disease (CAD), stroke, renal disease, and all-cause mortality. For every 7.5-mm Hg increase in diastolic blood pressure, CAD risk increases 29% and stroke risk increases 46%. These risks have been shown for women as well as for men. Even within the high-normal blood pressure range, higher measurements result in greater risk of cardiovascular diseases. (9-10) It has been reported that diet and nutritional supplements are effective in reducing elevated blood pressure and reducing the risk of heart attack and stroke. (11-15) Diet and supplements have also been shown to have effects in reducing blood cholesterol. (16, 17)

Traditional dietary control has focused on reducing intake of saturated fat and cholesterol. Recent studies have suggested that the traditional focus of lipid management may have been overly simplistic and that diets might be more effective if more attention was given on including certain foods or factors rather than just avoiding saturated fat and cholesterol. Gardner et al 2005 reported improved results with more plant-based foods, such as whole grains, vegetables, legumes, and fruits while simultaneously limiting saturated fat and cholesterol. (17) It has been reported that nutritional supplements and diet can reduce serum lipids and blood pressure. There are no reports on the effects of nutritional supplement on HRV despite the close link of the autonomic nervous system activity on regulation of blood pressure.

The Standard Process 21 day Purification Program consists of a controlled food intake regimen of mostly fruit and vegetables with restricted calories, protein and fats plus daily use of herbal and whole food based supplements. A recent case series of 28 chiropractic patients showed that the use of the SPPP resulted in significantly lowered total cholesterol. (18).

This study will investigate the effects of the SPPP in participants with elevated total cholesterol. The program requires the subjects to eat a modified; mostly fruits and vegetables diet and take the SPPP nutritional supplements for three weeks

The outcome measures of this study are supported in the literature as risk factors for cardiovascular and other conditions, e.g., serum lipids, C - reactive protein, homocystine, blood pressure, high BMI and heart rate variability (HRV).

ELIGIBILITY:
Inclusion Criteria:

* The two experimental groups will be 1. normal weight participants (BMI < 26) and 2. overweight participants (BMI 26 or above).
* All participants will have total cholesterol levels over 180.
* Both male and female subjects between the ages of 18-65 will be included in the study.

Exclusion Criteria:

* Exclusion criteria are based on factors that could interfere with the effects of the SPPP on the outcome measures and/or the safety of the participants as follows:
* Individuals with diabetes, heart, kidney, thyroid disorders, neurological diseases, and chronic disease will be excluded from the study.
* Female subjects who are pregnant or breast feeding and those using blood lipid modifying medications and/or supplements drugs and/or hypertension will be excluded from study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2008-07; Primary Completion 2009-03 (Estimated); Study Completion 2009-03 (Estimated)

PRIMARY OUTCOMES:
Serum lipids | Before and 3 weeks after starting SPPP (dietary modification + whole food supplements)

SECONDARY OUTCOMES:
Total cholesterol, LDL cholesterol, HDL cholesterol, triglycerides, homocysteine, C-reactive protein, blood pressure, heart rate variability, body mass index | Before and 3 weeks after starting SPPP (dietary modification + whole food supplements)

CONTACTS AND LOCATIONS:
Locations (1):
- Logan College of Chiropractic, Chesterfield, Missouri, United States